CLINICAL TRIAL: NCT00254423
Title: Therapy of Early Chronic Phase Chronic Myelogenous Leukemia (CML) With Dasatinib (BMS-354825)
Brief Title: Dasatinib in Treating Patients With Early Chronic Phase Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0422; NCI-2012-01317 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-2010-00440; 2005-0422 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2005-11-14; First posted 2005-11-16 (Estimated); Results first posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Chronic Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Philadelphia Chromosome Positive, BCR-ABL1 Positive Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dasatinib (Experimental): Patients receive dasatinib PO QD for up to 15-18 years.
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Given PO
  Other Names: BMS-354825; Dasatinib Hydrate; Dasatinib Monohydrate; Sprycel

SUMMARY:
The goal of this clinical research study is to learn if BMS-354825 (dasatinib) can help to control CML in chronic phase. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
Dasatinib is an anticancer drug that is designed to block the function of BCR-ABL, which is the abnormal protein responsible for causing leukemia in certain cells.

Before you can start therapy on this study, you will have what are called "screening tests." These tests will help the doctor decide if you are eligible to take part in the study. You will have a complete medical history and physical exam. Blood (about 2 tablespoons) will be collected for routine tests. You will also have a bone marrow biopsy and aspiration. To collect a bone marrow biopsy and aspiration, an area of the hip or chest bone is numbed with anesthetic and a small amount of bone marrow and bone is withdrawn through a large needle. Women who are able to have children must have a negative blood or urine pregnancy test. If you are found to be eligible to take part in this study and you agree, you will take dasatinib once every day while on study. Dasatinib should be taken by mouth with water.

Every 1-2 weeks during the first 4 weeks of the study, you will have around 2 tablespoons of blood drawn for routine blood tests. The blood tests will be repeated every 4-6 weeks until 1 year from when you started therapy and then every 3-4 months until 2 years, then as often as the doctor thinks it is needed. A bone marrow aspiration will also be taken to check the status of the disease every 3-4 months for the first year and then as often as the doctor thinks it is needed for as long as you are on the study.

You will be given a medication diary to monitor any missed doses. You will also be asked to visit the doctor for a physical exam and to have vital signs measured periodically. These visits will be scheduled at least every 3-4 months for the first year, then recommended every 6 to 12 months while you are on the study. The visits may be scheduled more often depending on the status of the disease.

Treatment may be continued for up to 8-10 years or as long as the doctor feels it is necessary to control the leukemia. If the disease gets worse or you experience any intolerable side effects, you will be taken off the study and your doctor will discuss other treatment options with you. If you decide to stop participating in the study, you are encouraged to discuss your decision with your study doctor.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Ph-positive or Bcr-Abl positive CML in early chronic phase CML (i.e., time from diagnosis </= 12 months). Except for hydroxyurea, patients must have received no or minimal prior therapy, defined as <1 month (30 days) of prior IFN-alpha (with or without ara-C) and/or an FDA approved TKI
* Continued from above #1: Clonal evolution defined as the presence of additional chromosomal abnormalities other than the Ph chromosome has been historically been included as a criterion for accelerated phase. However, patients with clonal evolution as the only criterion of accelerated phase have a significantly better prognosis, and when present at diagnosis may not impact the prognosis at all. Thus, patients with clonal evolution and no other criteria for accelerated phase will be eligible for this study
* Age >/= 16 years (Age >18 years to participate in optional symptom burden assessment)
* ECOG performance of 0-2
* Adequate end organ function, defined as the following: total bilirubin <1.5 x ULN, SGPT <2.5x ULN, creatinine <1.5x ULN
* Patients must sign an informed consent indicating they are aware of the investigational nature of this study, in keeping with the policies of the hospital.
* Reliable telephone access to receive calls from an interactive voice response system (IVR) (only applicable to patients who will participate in optional symptom burden assessment)

Exclusion Criteria:

* New York Heart Association (NYHA) cardiac class 3-4 heart disease
* Cardiac Symptoms: Patients meeting the following criteria are not eligible unless cleared by Cardiology: Uncontrolled angina within 3 months; Diagnosed or suspected congenital long QT syndrome; Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes); Prolonged QTc interval on pre-entry electrocardiogram (> 450 msec) on both the Fridericia and Bazett's correction; Uncontrolled hypertension; History of significant bleeding disorder unrelated to cancer, including:
* Cont: Diagnosed congenital bleeding disorders (von Willebrand's disease) Diagnosed acquired bleeding disorder w/in 1 year (acquired anti-factor VIII antibodies);Pts currently taking drugs that are generally accepted to have a risk of causing Torsades de Pointes including: quinidine, procainamide, disopyramide amiodarone, sotalol, ibutilide, dofetilide erythromycins, clarithromycin chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine.
* Patients with active, uncontrolled psychiatric disorders including: psychosis, major depression, and bipolar disorders
* Women of pregnancy potential must practice 2 effective methods of birth control during the course of the study, in a manner such that risk of failure is minimized.Prior to study enrollment, women of childbearing potential (WOCBP) must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
* Continued: Women must continue birth control for the duration of the trial and at least 3 months after the last dose of study drug; Pregnant or breast-feeding women are excluded; All WOCBP MUST have a negative pregnancy test prior to first receiving investigational product. If the pregnancy test is positive, the patient must not receive investigational product and must not be enrolled in the study.
* Patients in late chronic phase (i.e., time from diagnosis to treatment >12 months), accelerated or blast phase are excluded.
* The definitions of CML phases are as follows: a) Early chronic phase: time from diagnosis to therapy </= 12 months; Late chronic phase: time from diagnosis to therapy > 12 months, b) Blastic phase: presence of 30% blasts or more in the peripheral blood or bone marrow, c) Accelerated phase CML: presence of any of the following features: Peripheral or marrow blasts 15% or more, Peripheral or marrow basophils 20% or more, Thrombocytopenia < 100 x 10^9/L unrelated to therapy, Documented extramedullary blastic disease outside liver or spleen

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-11-08 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Masarova, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Jain P, Kantarjian H, Boddu PC, Nogueras-Gonzalez GM, Verstovsek S, Garcia-Manero G, Borthakur G, Sasaki K, Kadia TM, Sam P, Ahaneku H, O'Brien S, Estrov Z, Ravandi F, Jabbour E, Cortes JE. Analysis of cardiovascular and arteriothrombotic adverse events in chronic-phase CML patients after frontline TKIs. Blood Adv. 2019 Mar 26;3(6):851-861. doi: 10.1182/bloodadvances.2018025874. PMID 30885996
- [Derived] Issa GC, Kantarjian HM, Gonzalez GN, Borthakur G, Tang G, Wierda W, Sasaki K, Short NJ, Ravandi F, Kadia T, Patel K, Luthra R, Ferrajoli A, Garcia-Manero G, Rios MB, Dellasala S, Jabbour E, Cortes JE. Clonal chromosomal abnormalities appearing in Philadelphia chromosome-negative metaphases during CML treatment. Blood. 2017 Nov 9;130(19):2084-2091. doi: 10.1182/blood-2017-07-792143. Epub 2017 Aug 23. PMID 28835440
- [Derived] Jain P, Kantarjian H, Nazha A, O'Brien S, Jabbour E, Romo CG, Pierce S, Cardenas-Turanzas M, Verstovsek S, Borthakur G, Ravandi F, Quintas-Cardama A, Cortes J. Early responses predict better outcomes in patients with newly diagnosed chronic myeloid leukemia: results with four tyrosine kinase inhibitor modalities. Blood. 2013 Jun 13;121(24):4867-74. doi: 10.1182/blood-2013-03-490128. Epub 2013 Apr 25. PMID 23620574
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dasatinib
Started | 150
Completed | 150
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dasatinib
Number analyzed (Participants) | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 135
  >=65 years | 14
Age, Continuous [Median (Full Range); unit: years] | 48 [16 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 89
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 139
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 150

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Major Molecular Response at 12 Months
Description: Major Molecular Response (MMR) is BCR-ABL/ABL ratio </= 0.05
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 137
Participants | 103

2. Secondary Outcome: Overall Survival
Description: Time from date of treatment start until date of death due to any cause or last Follow-up.
Time Frame: Up to 19 years, 4 months and 6 days
Measure: Median (Full Range); unit: Months
Arm/Group | Dasatinib
Number analyzed (Participants) | 150
Months | NA [0.3 to 232] — OS median not reached due to insufficient number of participants with events

3. Secondary Outcome: Participants With Complete Cytogenic Response (CCR)
Description: Complete Cytogenic Response (CCR) is Ph positive 0%
Time Frame: Up to 19 years, 4 months and 6 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 150
Participants | 140

4. Secondary Outcome: Participants Who Developed the ABL Mutations
Description: ABL mutations will be assesses during treatment through Quanitiative PCR (qPCR) (RT-qPCR) or ABM mutational analysis using Sanger Sequencing or next-Generation Sequencing (NGS).
Time Frame: Up to 19 years, 4 months and 6 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 150
Participants | 7

ADVERSE EVENTS:
Time Frame: Up to 19 years, 4 months and 6 days
Arm/Group | Dasatinib
All-Cause Mortality (participants affected / at risk) | 4/150
Serious Adverse Events (participants affected / at risk) | 34/150
Other Adverse Events (participants affected / at risk) | 144/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib (N=150)
Abdominal Pain (General disorders) | 3 (3)
Allergic reaction (Immune system disorders) | 1 (1)
Allergy-Other : Angioedema/allergic reaction to Enalapril (Immune system disorders) | 1 (1)
Allergy-Other : Study drug (Dasatinib) overdose (Immune system disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Atrial Flutter (Cardiac disorders) | 1 (1)
Biventricular Heart Failure (Cardiac disorders) | 1 (1)
Cardiac ischemia/infarction (Cardiac disorders) | 2 (2)
Cardiac Pain (Cardiac disorders) | 1 (1)
Cellulitis (Infections and infestations) | 3 (5)
Chest Pain (General disorders) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 2 (3)
headache (Nervous system disorders) | 2 (2)
Infection (Infections and infestations) | 3 (3)
Left distal biceps tendon repair (Surgical and medical procedures) | 1 (1)
monoclonal gammopathy of undetermined significance (General disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neurology/Potential Drug Dependency (Nervous system disorders) | 1 (1)
Pain (General disorders) | 2 (3)
Back Pain (General disorders) | 1 (2)
Bone Pain (General disorders) | 1 (1)
Pancreatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 3 (4)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Prolonged QTc (Cardiac disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Squamous Cell Carcinoma of the skin -back of left ear (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous Cell Carcinoma of the Right Ear (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
unexpected pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib (N=150)
ACNE (Skin and subcutaneous tissue disorders) | 16 (20)
ALKALINE PHOSPHATASE (Metabolism and nutrition disorders) | 8 (9)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 8 (12)
ALLERGY/IMMUNOLOGY (OTHER) (Immune system disorders) | 8 (10)
ALOPECIA (Skin and subcutaneous tissue disorders) | 15 (16)
ALT SGPT (Investigations) | 15 (30)
ANEMIA (Blood and lymphatic system disorders) | 27 (33)
ANOREXIA (Metabolism and nutrition disorders) | 7 (7)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 8 (13)
AST SGOT (Investigations) | 25 (32)
AUDITORY/EAR (OTHER) (Ear and labyrinth disorders) | 8 (8)
BILIRUBIN (Investigations) | 8 (14)
BLURRED VISION (Eye disorders) | 33 (53)
CARDIAC ARRHYTHMIA (OTHER) (Cardiac disorders) | 7 (7)
CARDIAC GENERAL (OTHER) (Cardiac disorders) | 14 (18)
CHOLESTEROL (Investigations) | 7 (9)
CONSTIPATION (Gastrointestinal disorders) | 51 (92)
CONSTITUTIONAL SYMPTOMS (OTHER) (General disorders) | 31 (48)
COUGH (Respiratory, thoracic and mediastinal disorders) | 39 (52)
CREATININE (Investigations) | 9 (9)
DERMATOLOGY/SKIN (OTHER) (Skin and subcutaneous tissue disorders) | 34 (60)
DIARRHEA (Gastrointestinal disorders) | 88 (219)
DIZZINESS (Nervous system disorders) | 68 (138)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 83 (188)
EDEMA (General disorders) | 12 (17)
EDEMA: HEAD AND NECK (General disorders) | 19 (30)
EDEMA: LIMB (General disorders) | 44 (68)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 8 (11)
FATIGUE (General disorders) | 115 (269)
FEVER WITHOUT NEUTROPENIA (General disorders) | 47 (92)
FLUSHING (Vascular disorders) | 7 (8)
GASTROINTESTINAL (OTHER) (Gastrointestinal disorders) | 39 (61)
HEMOGLOBIN (Blood and lymphatic system disorders) | 34 (56)
HEMORRHOIDS (Gastrointestinal disorders) | 7 (7)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 19 (28)
HYPERKALEMIA (Metabolism and nutrition disorders) | 8 (9)
HYPERTENSION (Vascular disorders) | 23 (25)
HYPERURICEMIA (Metabolism and nutrition disorders) | 9 (11)
HYPOKALEMIA (Metabolism and nutrition disorders) | 7 (8)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 13 (15)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 7 (8)
INFECTION (Infections and infestations) | 7 (7)
INFECTION (OTHER) (Infections and infestations) | 22 (38)
INFECTION UNKNOWN ANC (SINUS) (Infections and infestations) | 8 (8)
INFECTION W NORMAL ANC (LUNG - PNEUMONIA) (Infections and infestations) | 8 (10)
INFECTION W NORMAL ANC (SINUS) (Infections and infestations) | 8 (12)
INFECTION W NORMAL ANC (URINARY TRACT NOS) (Infections and infestations) | 8 (9)
INFECTION WITHOUT NEUTROPENIA (Infections and infestations) | 10 (12)
INSOMNIA (Psychiatric disorders) | 24 (27)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 8 (8)
MEMORY IMPAIRMENT (Nervous system disorders) | 43 (65)
MENTAL STATUS (Nervous system disorders) | 7 (7)
METABOLIC/LABORATORY (OTHER) (Metabolism and nutrition disorders) | 13 (15)
MOOD ALTERATION (ANXIETY) (Psychiatric disorders) | 24 (25)
MOOD ALTERATION (DEPRESSION) (Psychiatric disorders) | 21 (28)
MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 7 (7)
MUSCULOSKELETAL (OTHER) (Musculoskeletal and connective tissue disorders) | 44 (63)
MYALGIA (Musculoskeletal and connective tissue disorders) | 11 (18)
NAUSEA (Gastrointestinal disorders) | 79 (163)
NEUROLOGY (OTHER) (Nervous system disorders) | 39 (69)
NEUROPATHY: MOTOR (Nervous system disorders) | 7 (11)
NEUROPATHY: SENSORY (Nervous system disorders) | 34 (71)
NEUTROPHILS (ANC/AGC) (Investigations) | 11 (17)
OCULAR VISUAL (OTHER) (Eye disorders) | 60 (130)
PAIN (ABDOMEN NOS) (Gastrointestinal disorders) | 22 (30)
PAIN (BACK) (Musculoskeletal and connective tissue disorders) | 23 (31)
PAIN (BONE) (Musculoskeletal and connective tissue disorders) | 24 (35)
PAIN (CHEST/THORAX) (General disorders) | 16 (17)
PAIN (EXTREMITY-LIMB) (General disorders) | 19 (24)
PAIN (HEAD/HEADACHE) (Nervous system disorders) | 72 (132)
PAIN (JOINT) (Musculoskeletal and connective tissue disorders) | 14 (16)
PAIN (MUSCLE) (General disorders) | 55 (101)
PAIN (ORAL CAVITY) (Gastrointestinal disorders) | 20 (37)
PAIN (OTHER) (General disorders) | 30 (51)
PAIN (THROAT/PHARYNX/LARYNX) (Respiratory, thoracic and mediastinal disorders) | 10 (10)
PALPITATIONS (Cardiac disorders) | 18 (26)
PERIORBITAL EDEMA (Eye disorders) | 20 (27)
PLATELETS (Investigations) | 33 (61)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 39 (72)
PRURITUS (Skin and subcutaneous tissue disorders) | 12 (18)
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 8 (12)
PULMONARY (OTHER) (General disorders) | 19 (20)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 45 (86)
RENAL/GENITOURINARY (OTHER) (Renal and urinary disorders) | 15 (17)
RIGORS/CHILLS (General disorders) | 12 (13)
SEXUAL/REPRODUCTIVE (OTHER) (Reproductive system and breast disorders) | 13 (14)
SINUS BRADYCARDIA (Cardiac disorders) | 11 (12)
SWEATING (General disorders) | 14 (14)
ULCERATION (General disorders) | 17 (21)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 10 (14)
URINARY FREQUENCY (Renal and urinary disorders) | 7 (8)
VOMITING (Gastrointestinal disorders) | 46 (94)
WATERY EYE (Eye disorders) | 29 (33)
WATERY EYES (Eye disorders) | 29 (40)
WEIGHT GAIN (Investigations) | 12 (13)
WEIGHT LOSS (Investigations) | 12 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/23/NCT00254423/Prot_SAP_001.pdf
  • Informed Consent Form (2020-03-05): https://cdn.clinicaltrials.gov/large-docs/23/NCT00254423/ICF_000.pdf